CLINICAL TRIAL: NCT06817499
Title: Treatment of Olfactory Dysfunction Using Vagus Nerve Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Lundström, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03779-01_s3; 2021-06527 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hyposmia
Keywords: VNS; Hyposmia; Olfaction; Olfaction Disorders; Sensation Disorders; Vagus Nerve
MeSH Terms: conditions — Anosmia; Olfaction Disorders; Sensation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olfactory training with nasal inserts + VNS (Experimental): Participants will complete olfactory training with scented nose plugs along with VNS
  Interventions: Other: Nasal Insert + VNS
- Olfactory training with nasal inserts only (Active Comparator): Participants will complete olfactory training with scented nose plugs
  Interventions: Other: Nasal Insert

INTERVENTIONS:
Other: Nasal Insert + VNS — Participants will complete olfactory training with scented nose plugs along with VNS
  Arms: Olfactory training with nasal inserts + VNS
Other: Nasal Insert — Participants will complete olfactory training with scented nose plugs
  Arms: Olfactory training with nasal inserts only

SUMMARY:
Hyposmia, a reduced sense of smell, is commonly linked to viral infections like COVID-19. Currently, the sole recommended treatment is olfactory training, a method that is both time-intensive and limited in its effectiveness. Our team has previously evaluated a new type of olfactory training using nasal inserts that show increased adherence to training (compared to standard olfactory training using common household odors) but with similar treatment effect. The investigators recently demonstrated that brief transcutaneous vagus nerve stimulation (VNS) in the cymba conchae region affected participants olfactory abilities but only when a stimulation frequency relevant to olfactory bulb processing frequencies was used. The notion that VNS might modulate olfactory functions stems from findings in rats where VNS of the cervical nerve inhibited neurons within the periglomerular layers of the olfactory bulb. Although there is no known monosynaptic connection between the vagus nerve and the olfactory system in humans, VNS activates areas with mono-synaptic connections to the olfactory bulb, such as amygdala, hippocampus, and the hypothalamus. Given that VNS modulates the olfactory bulb in rats and our treatment protocol modulate olfactory functions in humans, the investigators hypothesize that VNS, when paired with olfactory training, will enhance olfactory functions in patients with hyposmia.

DETAILED DESCRIPTION:
Participants with hyposmia will be recruited and randomly assigned to one of two treatment groups. One group will engage in olfactory training using nasal inserts while the other will use olfactory training with nasal inserts along with VNS. Both interventions will take place at home, Monday through Friday, over a two-month period. To evaluate the outcomes, subjective and objective measures of olfactory function will be collected before, during, and after the treatment, along with assessments of quality of life and overall well-being. Treatment adherence will also be evaluated at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Correct age (18-65)
* Physically and cognitively capable of participating in the study
* Having appropriate olfactory screening test scores (hyposmic)

Exclusion Criteria:

* History of heart conditions
* Individuals with other diagnoses that could affect the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Sniffin' Sticks TDI test (objective olfactory function) | From enrollment to the end of treatment at 8 weeks
  Objective olfactory function will be measured using the Sniffin' Sticks TDI extended test (Burghart Messtechnik) which gives separate scores for odor threshold, odor discrimination, and odor identification; as well as a summated score (TDI) of objective olfactory function.
Self rated olfaction questionnaire (subjective olfactory function) | From enrollment to the end of treatment at 8 weeks
  Does the use of VNS increase the effect of olfactory training on subjective qualitative (parosmia) and quantitative (hyposmia) symptoms compared to only olfactory training? For this outcome, we will use self-ratings of qualitative and quantitative olfactory function, for example "Do you experience smell distortion (parosmia)?" (if yes, rate your problem from 0 to 10) and "rate your sense of smell from 0 to 10"
General Wellbeing Questionnaire (general wellbeing) | From enrollment to the end of treatment at 8 weeks
  Does the use of VNS increase the effect of olfactory training on subjective general wellbeing compared to only olfactory training? For this outcome, we will use the General Wellbeing Questionnaire (GWB).
Adherence to training questionnaire (Compliance) | From enrollment to the end of treatment at 8 weeks
  Does the use of VNS affect the compliance of olfactory training compared to olfactory training only? For this outcome, we will use a questionnaire that participants answer during their final visit. The questionnaire separately assesses consistency, perceived tediousness, forgetfulness, and cause for potential discontinuation of the training, for example by asking "how many times did you forget your training?"

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
anonymized data